CLINICAL TRIAL: NCT04209686
Title: Phase 2 Study of Paclitaxel, Pembrolizumab and Olaparib in Previously Treated Advanced Gastric Adenocarcinoma
Brief Title: Paclitaxel, Pembrolizumab and Olaparib in Previously Treated Advanced Gastric Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J19135; IRB00209006 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Advanced Gastric Adenocarcinoma
Keywords: Paclitaxel; Olaparib; Pembrolizumab; Immunotherapy; Anti-PD-1; PARP inhibitors; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; olaparib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Measurable Disease (Experimental): All Participants will receive Paclitaxel, Olaparib and Pembrolizumab.
  Interventions: Drug: Paclitaxel; Drug: Olaparib; Drug: Pembrolizumab
- Arm 2: Cohort 2-Unmeasurable Disease (Experimental): All Participants will receive Paclitaxel, Olaparib and Pembrolizumab.
  Interventions: Drug: Paclitaxel; Drug: Olaparib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Paclitaxel — 1. Patients will receive treatment on Day 1 and 8 starting with cycle 2.
  2. Paclitaxel (80 mg) will be administered IV on days 1 and 8 starting with cycle 2 (every 21 days).
  3. Drug - Paclitaxel - 80mg IV
  Other Names: Taxol
Drug: Olaparib — 1. Olaparib will be taken by mouth daily for 3 weeks (every 21 days).
  2. Drug - 100 mg or 300mg
  Other Names: Lynparza
Drug: Pembrolizumab — 1. Patients will receive treatment every 21 days.
  2. Pembrolizumab (200 mg) will be administered IV on day 1 (every 21 days).
  3. Drug - 200mg IV
  Other Names: MK-3475; Keytruda

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of paclitaxel plus olaparib and pembrolizumab in patients with previously treated advanced Gastric Cancer (GC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Must have advanced gastric or gastroesophageal cancer.
* Must have received only one prior line of systemic therapy for advanced disease and experienced disease progression on this regimen..
* For Cohort 1: Must have the presence of measurable lesion.
* Must agree to have a biopsy.
* Life expectancy of greater than 3 months.
* Patients must have adequate organ and marrow function defined by study - specified laboratory tests.
* Woman of childbearing potential must have a negative pregnancy test.
* Must use acceptable form of birth control while on study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Require any antineoplastic therapy.
* Require any other form of systemic or localized antineoplastic therapy.
* Has received prior therapy with paclitaxel or PARP inhibitor. Previous paclitaxel may be allowed if no progression on or within 6 months of receiving this drug.
* Hypersensitivity reaction to any paclitaxel, pembrolizumab or related compounds and/or to any of the components.
* Allergy to dexamethasone, diphenhydramine and famotidine.
* Is taking a moderate or strong CYP3A inhibitor.
* Has uncontrolled intercurrent acute or chronic medical illness.
* Has a known additional malignancy that is progressing and has required active treatment within the past 1 year.
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to study treatment.
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is currently or has participated in another investigational study within 4 weeks prior to receiving study drug.
* Has an active known or suspected autoimmune disease.
* Has a diagnosis of immunodeficiency.
* Prior tissue or organ allograft or allogeneic bone marrow transplantation.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. .
* Requires daily supplemental oxygen.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
* Infection with HIV or hepatitis B or C at screening.
* Has uncontrolled infection requiring systemic therapy..
* Subjects unable to undergo venipuncture and/or tolerate venous access.
* Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Woman who are pregnant or breastfeeding.
* A woman of childbearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to study drug initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 4 years
  OS will be measured from the date of first dose until death or end of follow-up. All subjects who receive at least one dose of the 3-drug combination will be included. Subjects who discontinue treatment prior to Cycle 2 will not be included in the analysis. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which that patient was known to be alive. Estimation based on the Kaplan-Meier curve.

SECONDARY OUTCOMES:
The number of patients experiencing study drug-related toxicities. | 4 years
  Number of participants experiencing drug-related adverse events requiring treatment discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bever, MD, Principal Investigator — Johns Hopkins Medical Institution
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No